CLINICAL TRIAL: NCT02899455
Title: Efficacy and Safety of Co-administered HGP0904, HGP0608 and HGP0816 in Patients With Hypertension and Dyslipidemia: A Randomized, Double-blind, Multicenter, Phase 3 Study
Brief Title: Clinical Efficacy and Safety Evaluation of Co-administered HGP0904, HGP0608 and HGP0816 in Patients With Hypertension and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALRO-301
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental (Experimental): HGP0904 + HGP0608 + HGP0816, once daily
  Interventions: Drug: HGP0904; Drug: HGP0608; Drug: HGP0816
- Active Comparator1 (Active Comparator): HGP0904 placebo + HGP0608 + HGP0816, once daily
  Interventions: Drug: HGP0608; Drug: HGP0816; Drug: HGP0904 Placebo
- Active Comparator2 (Active Comparator): HGP0904 + HGP0608 + HGP0816 placebo, once daily
  Interventions: Drug: HGP0904; Drug: HGP0608; Drug: HGP0816 Placebo

INTERVENTIONS:
Drug: HGP0904
  Arms: Active Comparator2; Experimental
Drug: HGP0608
Drug: HGP0816
  Arms: Active Comparator1; Experimental
Drug: HGP0904 Placebo
  Arms: Active Comparator1
Drug: HGP0816 Placebo
  Arms: Active Comparator2

SUMMARY:
A phase 3 study to evaluate efficacy and safety of Co-administered HGP0904, HGP0608 and HGP0816 in Patients with Hypertension and Dyslipidemia

DETAILED DESCRIPTION:
This study is designed as a multi-center, double-blinded, randomized, phase 3 clinical trial to evaluate the efficacy and safety of Co-administered HGP0904, HGP0608 and HGP0816 in Patients with Hypertension and Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

1. 19 ≤ age ≤ 75
2. at Visit 1 1) BP: sitDBP ≥ 90mmHg 2) Cholesterol : LDL-C ≤ 250mg/dL, TG < 400mg/dL
3. at Visit 2 : after TLC (after 4weeks) 1) BP: 80 mmHg ≤ sitDBP < 110mmHg 2) Cholesterol : following risk category (Cardiovascular Risk category) A : CHD risk factor 0 - 1, 160mg/dL ≤ LDL-C ≤ 250mg/dL B①: CHD risk factor≥2 and 10 year risk <10%, 160mg/dL ≤ LDL-C ≤ 250mg/dL B②: CHD risk factor≥2 and 10 year risk =10-20%, 130mg/dL ≤ LDL-C ≤ 250mg/dL C : CHD/CHD risk equivalents* or 10 year risk>20 ,100mg/dL ≤ LDL-C ≤ 250mg/dL 3) TG < 400mg/dL 4. Patients understood the contents and purpose of this trial and signed informed consent form

Exclusion Criteria:

1. At Visit 1, BP difference SBP ≥20mmHg or DBP ≥10mmHg
2. Tolerance or Hypersensitivity Angiotensin II receptor blocker or HMG-CoA. reductase inhibitor, Calcium channel blocker(dihydropyridine) or Multi-drug allergy
3. Fibromyalgia, myopathy, rhabdomyolysis or acute myopathy or medical history of adverse effect to statin
4. CPK normal range ≥ 3times
5. Uncontrolled primary hypothyroidism(TSH normal range ≥ 2 times)
6. Renal disease or suspected renal disease (Scr ≥ 2mg/dL, AST or ALT≥2 times)
7. Active gout or hyperuricemia(at Visit 1, uric acid > 9mg/dL)
8. IDDM or uncontrolled diabetes mellitus (HbA1c>9%)
9. ventricular arrhythmia
10. medical history

    * severe cerebrovascular disease within 6 months (cerebral infarction, cerebral hemorrhage), hypertension
    * encephalopathy, transient cerebral ischemic attack(TIA)
    * severe heart disease(heart failure of NYHA class III-IV), valvular disease of heart or myocardial infarction and unstable angina
    * angioplasty or coronary artery bypass graft(CABG) surgery within 6months

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in LDL-cholesterol at Week 8 | baseline and 8 weeks
Change from baseline in sitDBP at Week 8 | baseline and 8 weeks

SECONDARY OUTCOMES:
Percentage change from baseline in LDL cholesterol at Week 4 | baseline and 4 weeks
Percentage change from baseline in Total cholesterol, HDL cholesterol, Triglyceride at Week 4,8 | baseline, 4weeks and 8 weeks
Change from baseline in sitDBP at Week 4 | baseline and 4weeks
Change from baseline in sitSBP at week 4, 8 | baseline, 4weeks and 8 weeks
Proportion of subjects achieving LDL-cholesterol goals by cardiovascular risk category at Week 4, 8 | baseline, 4weeks and 8 weeks
Proportion of subjects achieving Blood Pressure control by cardiovascular risk category at Week 4, 8 | baseline, 4weeks and 8 weeks
Proportion of subjects achieving LDL-cholesterol goals and Blood Pressure control by cardiovascular risk category at Week 4, 8 | baseline, 4weeks and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 23 institutions including Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HY, Kim SY, Choi KJ, Yoo BS, Cha DH, Jung HO, Ryu DR, Choi JH, Lee KJ, Park TH, Oh JH, Kim SM, Choi JY, Kim KH, Shim J, Kim WS, Choi SW, Park DG, Song PS, Hong TJ, Rhee MY, Rha SW, Park SW. A Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and the Tolerability of a Triple Combination of Amlodipine/Losartan/Rosuvastatin in Patients With Comorbid Essential Hypertension and Hyperlipidemia. Clin Ther. 2017 Dec;39(12):2366-2379. doi: 10.1016/j.clinthera.2017.10.013. Epub 2017 Nov 14. PMID 29150250